CLINICAL TRIAL: NCT03151148
Title: A First in Man Evaluation of the Safety and Efficacy of an Allogeneic Targeted Microbiome Transplant in Adults With Moderate-to-Severe Atopic Dermatitis (ADRN-08)
Brief Title: Targeted Microbiome Transplant in Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ADRN-08
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Results first posted 2020-05-22 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Atopic Dermatitis (AD)
Keywords: allogeneic targeted microbiome transplant (TMT); dysbiosis in AD; Staphylococcus aureus colonized skin; antimicrobial peptides (AMPs); randomized trial
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Trail Making Test

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TMT Lotion (Experimental): The targeted microbiome transplant (TMT) lotion will be provided in single-dose sealed packets. The lotion should be stored at 4°Celsius (=39.2 degrees Fahrenheit). Participants randomized to active TMT will apply 2 grams of TMT to each ventral aspect of their arm (wrist to upper humerus). Frequency of lotion application: topical application administered twice daily for one week.
  Interventions: Biological: TMT Lotion
- Placebo Lotion (Placebo Comparator): Placebo lotion will be provided in single-dose sealed packets. The lotion should be stored at 4°Celsius (=39.2 degrees Fahrenheit). Participants randomized to placebo will apply 2 grams of placebo to each ventral aspect of their arm (wrist to upper humerus). Frequency of lotion application: topical application administered twice daily for one week.
  Interventions: Drug: Placebo Lotion

INTERVENTIONS:
Biological: TMT Lotion — TMT product and Vegetable glycerin-Cetaphil®
  Other Names: Targeted Microbiome Transplant (TMT) Lotion
  Arms: TMT Lotion
Drug: Placebo Lotion — Cetaphil® moisturizing lotion and vegetable glycerin
  Other Names: Placebo for Targeted Microbiome Transplant (TMT) Lotion
  Arms: Placebo Lotion

SUMMARY:
The purpose of this study is to examine the safety and effectiveness of a new therapy, commensal lotion containing infection fighting bacteria, on decreasing or eliminating the infection causing bacteria found on the skin of Atopic Dermatitis (AD) patients.

DETAILED DESCRIPTION:
This study will enroll adult participants, 18-60 years of age, with moderate-to-severe atopic dermatitis (AD) and a positive Staphylococcus aureus (S. aureus) colonized lesion (at least 15 cm^2 in size) on the upper extremities.

Participants who are eligible based on their positive Staph culture results will be randomized to one of two treatments: Targeted Microbiome Transplant Lotion (TMT) or Placebo (2:1 randomization). One lesional site measuring at least 15 cm^2 and one non-lesional site of equal size will be identified on the participant's ventral upper extremities as the target swabbing areas. These sites will be photographed and marked for swabbing for reference at the participant's future visits. Participants will be instructed to apply investigational product with gloved hands to their ventral upper extremities bilaterally from the wrist to the upper humerus, which will include the identified lesional and non-lesional swabbing sites twice a day for 1 week starting on Day 0. Participants will return to clinic on Day 4 for the assessment of adverse events, the collection of skin swabs from the identified target sites, and to obtain additional investigational product and gloves. Participants will complete an additional clinic visit on Day 7 to correspond with the end of their 1 week treatment. During this visit, participants will be assessed for AEs and provide skin swab samples. All unused product and empty packets will be returned during the Day 4 and Day 7 visits. Three additional clinic visits on Days 8, 9, and 11 will be scheduled for additional skin swabs to assess the safety and the stability of the microbiome transplant and time to recurrence of Staph colonization. Participants will be followed through Day 38 to assess for safety and disease status.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

* Participant must be able to understand and provide informed consent;
* Fulfills the Atopic Dermatitis Research Network (ADRN) Standard Diagnostic Criteria (Appendix A) for active Atopic Dermatitis (AD);
* A Staphylococcus aureus (S. aureus) positive culture colonized lesion, at least 15 cm^2 in size, located on a ventral upper extremity (e.g., arm);
* An Investigator Global Assessment (IGA) score, on the ventral arms, of at least moderate severity;
* A body surface area (BSA), as measured by Mosteller BSA Calculator, between 1.26 m^2 (e.g., 4 feet, 10 inches and 85 pounds [38.6 Kg] and 2.25 m^2 (e.g., 6 feet, 3 inches and 210 pounds [95.5 Kg]; and
* Females of childbearing potential who are willing to use adequate contraception 30 days prior to the Screening Visit and until participation in the study is complete.

  --Females of childbearing potential must agree to use an acceptable method of birth control (e.g. total abstinence, oral contraceptives, intrauterine device [IUD], barrier method with spermicide, surgical sterilization or surgically sterilized partner, Depo-Provera, Norplant, NuvaRing, or hormonal implants) for the duration of study participation.
* Male participants who are willing to use an acceptable method of contraception (e.g. barrier methods with spermicide, surgical sterilization or surgically sterilized partner) or practice abstinence until participation in the study is complete.

Exclusion Criteria:

* Inability or unwillingness of participant to give written informed consent or comply with study protocol;
* Pregnant or lactating females, or females who desire to become pregnant and/or breast feed within the duration of study participation;
* Active bacterial, viral, or fungal skin infections;
* Any noticeable breaks or cracks in the skin on the upper extremities, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection;
* Sensitivity to or difficulty tolerating Dove fragrance-free bar soap, Cetaphil(R) Lotion, alcohol-based cleaners, macadamia nuts, soy, Vegetable glycerin, or palm kernels;
* Participants with prosthetic heart valves, pacemakers, intravascular catheters, or other foreign or prosthetic devices;
* Participants with Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier;
* Any participant who is immunocompromised (e.g. history of lymphoma, Human Immunodeficiency Virus (HIV)/ Acquired Immune Deficiency Syndrome (AIDS), Wiskott-Aldrich Syndrome) or has a history of malignant disease (with the exception of non-melanoma skin cancer);
* Participants with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol;
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study;
* Ongoing participation in another investigational trial or use of investigational drugs within 8 weeks, or 5 half-lives (if known), whichever is longer, of the Screening Visit;
* Treatment with biologics within 16 weeks of Screening Visit;
* Participants with close contacts (e.g. spouses, children, or members in the same household) that have severe barrier defects or are immunocompromised;
* Use of topical (including steroids and calcineurin inhibitors) Atopic Dermatitis (AD) treatments within 7 days of the Treatment Visit; Use of topical steroids on areas outside of where investigational product is to be applied may be permitted, per investigator discretion;
* Treatment of AD with prescription moisturizers classified as medical device (e.g., Atopiclair®, MimyX®, Epicerum®, Cerave®, etc.) within 7 days of the Treatment Visit;
* Use of any oral or topical antibiotics within 7 days of the Treatment Visit;
* Participants who have taken a bleach bath within 7 days of the Treatment Visit;
* Use of any oral AD therapies (antihistamines, steroids, immunosuppressive therapies) within 28 days of the Treatment Visit; or
* Any phototherapy for skin disease (such as narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + UVA [PUVA]) or regular use (more than 2 visits per week) of a tanning bed within 28 days of the Treatment Visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gallo, M.D., Ph.D., Study Chair — University of California, San Diego: Dermatology Clinical Trials Unit
Locations (2):
- United States (2):
  - University of California - San Diego, San Diego, California
  - National Jewish Health General Clinical Research Center, Denver, Colorado

REFERENCES:
- [Derived] Nakatsuji T, Hata TR, Tong Y, Cheng JY, Shafiq F, Butcher AM, Salem SS, Brinton SL, Rudman Spergel AK, Johnson K, Jepson B, Calatroni A, David G, Ramirez-Gama M, Taylor P, Leung DYM, Gallo RL. Development of a human skin commensal microbe for bacteriotherapy of atopic dermatitis and use in a phase 1 randomized clinical trial. Nat Med. 2021 Apr;27(4):700-709. doi: 10.1038/s41591-021-01256-2. Epub 2021 Feb 22. PMID 33619370
- See also: National Institute of Allergy and Infectious Disease (NIAID) Website — http://www.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of patients with active atopic dermatitis took place between 20 September 2017 through 24 April 2019 at 2 clinical centers in the US: National Jewish Health: Division of Pediatric Allergy and Clinical Immunology and University of California - San Diego
Pre-assignment Details: Screened S. aureus positive participants requiring medication/therapy washout of ≤14 days to meet inclusion/exclusion criteria were randomized within 14 days of screening. Screened S. aureus positive participants requiring medication/therapy washout > 14 days, completed a Repeat Culture Visit after a washout, to confirm S. aureus colonization.
Groups:
- TMT Lotion: The targeted microbiome transplant (TMT) lotion was provided in single-dose sealed packets.
  Participants applied 2 grams of TMT to each ventral aspect of their arm (wrist to upper humerus). Frequency of lotion application: topical application administered twice daily for one week.
- Placebo Lotion: Placebo lotion was provided in single-dose sealed packets.
  Participants applied 2 grams of placebo to each ventral aspect of their arm (wrist to upper humerus). Frequency of lotion application: topical application administered twice daily for one week.
Period: Overall Study
Arm/Group | TMT Lotion | Placebo Lotion
Started | 36 | 18
Completed | 34 | 18
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants randomized and received at least one treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | TMT Lotion | Placebo Lotion | Total
Number analyzed (Participants) | 36 | 18 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 35 | 17 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Age Continuous (years)] | 29.4 (12.16) | 26.6 (10.18) | 28.4 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 19 | 6 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 29 | 15 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 15 | 8 | 23
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 18 | 54
Screening Staphylococcus aureus (S. aureus) blood agar growth score [Count of Participants; unit: Participants] — Measure of S. aureus colonies present on the participant's lesional skin, as measured by bacteria growth on a blood agar plate. A skin swab sample was collected from an area of lesional skin on the participant's upper extremity at their Screening Visit. Growth was measured as 0-4, increasing in relation to the amount of S. aureus present on the blood agar plate. In order to enroll, participants needed a positive S. aureus colonized lesion, with a growth score of at least 1.
  Participants
    1 | 11 | 5 | 16
    2 | 9 | 3 | 12
    3 | 5 | 2 | 7
    4 | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Per-Participant Daily Event Rate: Serious and Non-Serious Treatment Emergent Adverse Events (TEAEs)
Description: Per-participant daily event rate of TEAEs was calculated as the number of events per-participant-days at risk. Statistical method employed: Poisson generalized linear model with a log link function and including the natural log of the number of days active in the study during Day 0 to Day 8.
Time Frame: Day 0 to Day 8
Population: Safety sample: All participants who were randomized and received any doses of their assigned intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: events per-participant-day
Groups:
- Targeted Microbiome Transplant (TMT): The targeted microbiome transplant (TMT) lotion was provided in single-dose sealed packets.
  Participants applied 2 grams of TMT to each ventral aspect of their arm (wrist to upper humerus). Frequency of lotion application: topical application administered twice daily for one week.
Arm/Group | Targeted Microbiome Transplant (TMT) | Placebo Lotion
Number analyzed (Participants) | 36 | 18
events per-participant-day | 0.19 [0.12 to 0.29] | 0.34 [0.20 to 0.58]
Statistical Analysis 1: Comparison: Targeted Microbiome Transplant (TMT) vs Placebo Lotion; Test type: Superiority; p = 0.075, Negative Binomial Regression; Negative binomial generalized linear model, adjusting for site, offset by follow-up days within the outcome measure time frame; Risk Ratio (RR) = 0.56, 95% CI 2-sided [0.29 to 1.06] — TMT represents the numerator, placebo represents the denominator

2. Secondary Outcome: The Occurrence of at Least One Serious or Non-Serious Treatment Emergent Adverse Event (TEAE)
Description: The number of participants for which at least one treatment emergent adverse event (AE), defined as an increase in grade from baseline or from the last post-baseline value that does not meet grading criteria, was reported during the measure time frame.
Time Frame: Day 0 (after initiation of study treatment) through Day 8 (last day of study treatment)
Population: Safety sample: All participants who were randomized and received any doses of their assigned intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 36 | 18
Participants | 20 | 15
Statistical Analysis 1: Comparison: TMT Lotion vs Placebo Lotion; Test type: Superiority; p = 0.044, Chi-squared; Risk Difference (RD) = -0.28, 95% CI 2-sided [-0.51 to -0.04] — 95% exact unconditional confidence interval is based on the Santner and Snell method

3. Secondary Outcome: Per-Participant Daily Event Rate of Serious and Non-Serious Adverse Events (AEs)
Description: Per-participant daily event rate of serious and non-serious AEs was calculated by the number of events per-participant days active in the study during Screening to Day 38.
Time Frame: Screening (up to 38 days before initiation of treatment) to Day 38 (last day of study participation)
Population: Safety sample (all participants who are randomized and receive any amount of study drug)
Measure: Least Squares Mean (95% Confidence Interval); unit: events per-participant-day
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 36 | 18
events per-participant-day | 0.06 [0.04 to 0.09] | 0.09 [0.06 to 0.15]
Statistical Analysis 1: Comparison: TMT Lotion vs Placebo Lotion; Test type: Superiority; p = 0.121, Negative Binomial Regression; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.63, 95% CI 2-sided [0.36 to 1.13] — TMT represents the numerator, placebo represents the denominator

4. Secondary Outcome: The Occurrence of at Least One Serious or Non-Serious Adverse Event (AE)
Description: The number of participants for which at least one adverse event (AE) was reported
Time Frame: Screening (up to 38 days before initiation of treatment) to Day 38 (last day of study participation)
Population: Safety sample (all participants who are randomized and receive any amount of study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 36 | 18
Participants | 23 | 16
Statistical Analysis 1: Comparison: TMT Lotion vs Placebo Lotion; Test type: Superiority; p = 0.053, Chi-squared; Risk Difference (RD) = -0.25, 95% CI 2-sided [-0.46 to -0.04] — 95% exact unconditional confidence interval is based on the Santner and Snell method

5. Secondary Outcome: The Eczema Area and Severity Index (EASI) Score of the Ventral Arms at Specific Days During the Measure Time Frame
Description: The eczema area and severity index (EASI) for the ventral arms is a composite score measuring physical signs of atopic dermatitis. The scale ranges from 0-18. The components measuring severity are four signs/symptoms of atopic dermatitis: erythema, papulation, excoriation, and lichenification each scored on a scale of 0 (absent) to 3 (severe) for the ventral arms. The component measuring area is the percent area of the ventral arms with atopic dermatitis lesions scored on a scale of 0 (0%) to 6 (90-100%).
Time Frame: Days 0, 4, 7, 8 and 11
Population: Modified Intention-to-Treat (MITT) sample includes all randomized participants who provided skin swabs on Day 0 and Day 7 and administered 75 percent of doses of the study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
units on a scale
  Day 0 | 2.5 (1.47) | 2.2 (1.06)
  Day 4 | 2.5 (1.6) | 2.2 (0.98)
  Day 7 | 2.2 (1.51) | 1.9 (1.11)
  Day 8: number analyzed (Participants) | 34 | 15
  Day 8 | 2.1 (1.5) | 1.9 (1.14)
  Day 11 | 2.0 (1.47) | 1.7 (1.16)

6. Secondary Outcome: The Scoring Atopic Dermatitis (SCORAD) Score at Specific Days During the Measure Time Frame
Description: SCORAD (Severity scoring of Atopic Dermatitis) is a composite severity index comprising A) the amount/extent of body surface area affected; A= 0-100%, B) disease intensity assessed as sum of scores for 6 parameters (erythema, edema/papulation, oozing/crusting, excoriation, lichenification, and dryness), each graded from 0 (none) to 3 (severe); B= 0-18, and C) subjective symptom visual analog assessments for pruritus [0 (no itch) to 10 (worst imaginable itch)] and sleep loss [0 (no sleep loss) to 10 (worst imaginable sleep loss)] summed for a total symptom score; C=0-20. The SCORAD = A/5 + 7B/2 + C and ranges from 0 (no AD present) to 103 (severe).
Time Frame: Days 0, 4, 7, 8 and 11
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
units on a scale
  Day 0 | 50.0 (12.82) | 46.5 (12.76)
  Day 4 | 48.9 (13.48) | 45.5 (11.49)
  Day 7 | 43.8 (13.75) | 40.7 (12.96)
  Day 8: number analyzed (Participants) | 34 | 15
  Day 8 | 42.4 (13.45) | 43.3 (14.71)
  Day 11 | 40.5 (14.94) | 39.4 (15.13)

7. Secondary Outcome: The Rajka-Langeland (RL) Score at Specific Days During the Measure Time Frame
Description: The Rajka & Langeland (RL) eczema severity score is a simple assessment of AD severity as well as the classification of AD into mild, moderate, or severe. The score is based on the grading of: (i) eczema extent based on % body area affected, (ii) eczema course based on the number of months with remission during the previous year, and (iii) eczema intensity expressed in terms of nocturnal sleep disturbance due to itch. Each parameter is scored on a scale from 1-3, and the scores are summed. The RL score ranges from 3 to 9 (mild, 3-4; moderate, 4.5-7.5; severe, 8-9)
Time Frame: Days 0 and 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
units on a scale
  Day 0 | 7.0 (1.52) | 6.6 (1.41)
  Day 7 | 6.8 (1.59) | 6.5 (1.50)

8. Secondary Outcome: The Pruritus Visual Analog Scale (VAS) Score of the Ventral Arms at Specific Days During the Measure Time Frame
Description: The pruritus visual analog scale (VAS) asks participants to rate the status of their Pruritus based on the severity of their itch. Scores range from 0 to 10 (0 = no itch, 10 = worst imaginable itch)
Time Frame: Days 0, 4, 7, 8 and 11
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
units on a scale
  Day 0 | 6.1 (2.26) | 5.3 (2.59)
  Day 4 | 5.7 (2.44) | 4.7 (2.56)
  Day 7 | 4.2 (2.46) | 3.4 (2.40)
  Day 8: number analyzed (Participants) | 34 | 15
  Day 8 | 3.3 (2.08) | 3.3 (2.66)
  Day 11 | 3.2 (2.38) | 2.9 (2.66)

9. Secondary Outcome: The Abundance of Coagulase Negative Staphylococcal (CoNS) Species, as Measured by Culture, on Lesional and Non-Lesional Skin Within Each Treatment Group
Description: Amount of CoNS present on lesional and non-lesional skin measured by Colony Forming Units per centimeter squared (CFU/cm^2)
Time Frame: Days 0, 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: CFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
CFU/cm^2
  Day 0 - Lesional | 113.8 [31.45 to 411.48] | 81.8 [12.94 to 517.14]
  Day 0 - Non-lesional | 41.2 [11.40 to 149.23] | 78.8 [12.47 to 498.41]
  Day 4 - Lesional | 549.7 [151.99 to 1988.39] | 557.3 [88.14 to 3522.99]
  Day 4 - Non-lesional | 1351.5 [373.52 to 4890.38] | 16.5 [2.60 to 104.03]
  Day 7 - Lesional | 2421.9 [669.60 to 8759.87] | 335.2 [53.02 to 2118.99]
  Day 7 - Non-lesional | 2363.5 [653.20 to 8552.23] | 28.0 [4.43 to 176.98]
  Day 8 - Lesional | 371.0 [100.72 to 1366.65] | 19.2 [2.69 to 136.36]
  Day 8 - Non-lesional | 107.8 [29.27 to 397.34] | 20.6 [2.90 to 146.77]
  Day 11 - Lesional | 173.0 [47.83 to 625.77] | 15.6 [2.47 to 98.74]
  Day 11 - Non-Lesional | 102.0 [28.20 to 369.23] | 8.8 [1.39 to 55.36]
Statistical Analysis 1: Comparison: TMT Lotion; Lesional vs. Non-lesional within TMT at Day 0 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.261, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.76, 95% CI 2-sided [0.469 to 16.226] — All reported statistics are back-transformed into the original units of measurement. Baseline is defined as the pre-dose value at treatment initiation/Day 0. Lesional represents the numerator and Non-Lesional the denominator
Statistical Analysis 2: Comparison: TMT Lotion; Lesional vs. Non-lesional within TMT at Day 4 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.319, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.41, 95% CI 2-sided [0.069 to 2.393] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion; Lesional vs. Non-lesional within TMT at Day 7 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.978, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.02, 95% CI 2-sided [0.174 to 6.027] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion; Lesional vs. Non-lesional within TMT at Day 8 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.177, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.44, 95% CI 2-sided [0.570 to 20.749] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion; Lesional vs. Non-lesional within TMT at Day 11 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.558, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.70, 95% CI 2-sided [0.288 to 9.973] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Placebo Lotion; Lesional vs. Non-lesional within Placebo at Day 0 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.977, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.04, 95% CI 2-sided [0.082 to 13.151] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Placebo Lotion; Lesional vs. Non-lesional within Placebo at Day 4 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.007, Mixed Models Analysis; Geometric mean ratio (GMR) = 33.86, 95% CI 2-sided [2.672 to 429.219] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Placebo Lotion; Lesional vs. Non-lesional within Placebo at Day 7 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.055, Mixed Models Analysis; Geometric mean ratio (GMR) = 11.97, 95% CI 2-sided [0.945 to 151.752] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Placebo Lotion; Lesional vs. Non-lesional within Placebo at Day 8 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.957, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.93, 95% CI 2-sided [0.062 to 13.875] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Placebo Lotion; Lesional vs. Non-lesional within Placebo at Day 11 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.654, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.78, 95% CI 2-sided [0.141 to 22.607] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: The Abundance of Coagulase Negative Staphylococcal (CoNS) Species, as Measured by qPCR (Quantitative Polymerase Chain Reaction), on Lesional and Non-Lesional Skin Within Each Treatment Group
Description: Amount of CoNS on lesional and non-lesional skin measured by qPCR relative colony forming units per centimeter squared [rCFU/cm^2]
Time Frame: At days 0, 4, 7, 8 and 11
Population: Data were not collected.
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: The Change From Baseline Levels of Coagulase Negative Staphylococcal (CoNS) Bacteria Abundance, as Measured by Culture, on Lesional and Non-Lesional Skin Within Each Treatment Group
Description: as for outcome 9
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: CFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
CFU/cm^2
  Day 0 - Lesional | 3349.24 [564.555 to 19869.455] | 0.93 [0.072 to 11.936]
  Day 0 - Non-lesional | 1230.53 [207.421 to 7300.167] | 2.00 [0.155 to 25.694]
  Day 4 - Lesional | 4.83 [0.815 to 28.668] | 6.81 [0.529 to 87.659]
  Day 4 - Non-lesional | 32.77 [5.524 to 194.418] | 0.21 [0.016 to 2.686]
  Day 7 - Lesional | 21.29 [3.588 to 126.296] | 4.10 [0.318 to 52.725]
  Day 7 - Non-lesional | 57.31 [9.660 to 339.995] | 0.36 [0.028 to 4.569]
  Day 8 - Lesional | 3.26 [0.542 to 16.609] | 0.23 [0.017 to 3.286]
  Day 8 - Non-lesional | 2.61 [0.435 to 15.723] | 0.26 [0.019 to 3.670]
  Day 11 - Lesional | 1.52 [0.256 to 9.022] | 0.19 [0.015 to 2.457]
  Day 11 - Non-Lesional | 2.47 [0.417 to 14.679] | 0.11 [0.009 to 1.429]
Statistical Analysis 1: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.432, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.722, 95% CI 2-sided [0.2227 to 33.2594] — All reported statistics are back-transformed into the original units of measurement. Change from baseline is based on the difference in log10 post-baseline and log10 baseline values. Lesional represents the numerator and Non-Lesional the denominator
Statistical Analysis 2: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.133, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.147, 95% CI 2-sided [0.0121 to 1.8018] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.437, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.371, 95% CI 2-sided [0.0304 to 4.5392] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.863, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.247, 95% CI 2-sided [0.1002 to 15.5231] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.702, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.615, 95% CI 2-sided [0.0503 to 7.5106] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.675, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.465, 95% CI 2-sided [0.0128 to 16.8576] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.057, Mixed Models Analysis; Geometric mean ratio (GMR) = 32.638, 95% CI 2-sided [0.8994 to 1184.4298] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.181, Mixed Models Analysis; Geometric mean ratio (GMR) = 11.539, 95% CI 2-sided [0.3180 to 418.7586] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 9]; Test type: Superiority; p = 0.953, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.895, 95% CI 2-sided [0.0219 to 36.5559] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 10]; Test type: Superiority; p = 0.767, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.719, 95% CI 2-sided [0.0474 to 62.3828] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: The Change From Baseline Levels of Coagulase-Negative Staphylococcus (CoNS) Bacteria Abundance, as Measured by qPCR (Quantitative Polymerase Chain Reaction), on Lesional and Non-Lesional Skin Within Each Treatment Group
Description: Amount of CoNS present on lesional and non-lesional skin measured by qPCR (relative colony forming units per centimeter squared [rCFU/cm^2])
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: Data were not collected.
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: The Change From Baseline Levels of S. Hominis A9 Bacteria Abundance, as Measured by Quantitative Polymerase Chain Reaction (qPCR), on Lesional and Non-Lesional Skin Within Each Treatment Group
Description: Amount of S. hominis A9 present on lesional and non-lesional skin measured by qPCR (relative colony forming units per centimeter squared [rCFU/cm^2])
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: rCFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
rCFU/cm^2
  Day 0 - Lesional | 9802.91 [4635.353 to 20731.332] | 0.95 [0.325 to 2.785]
  Day 0 - Non-lesional | 7027.89 [3304.917 to 14944.772] | 0.43 [0.145 to 1.248]
  Day 4 - Lesional | 10620.64 [5022.021 to 22460.681] | 1.43 [0.488 to 4.182]
  Day 4 - Non-lesional | 3761.96 [1778.861 to 7955.848] | 0.72 [0.247 to 2.116]
  Day 7 - Lesional | 9986.58 [4722.202 to 21119.759] | 1.46 [0.500 to 4.286]
  Day 7 - Non-lesional | 4807.31 [2273.159 to 10166.564] | 0.79 [0.269 to 2.305]
  Day 8 - Lesional | 691.01 [324.818 to 1470.024] | 2.31 [0.745 to 7.188]
  Day 8 - Non-lesional | 875.33 [411.460 to 1862.155] | 0.62 [0.205 to 1.896]
  Day 11 - Lesional | 33.44 [15.813 to 70.721] | 2.15 [0.723 to 6.417]
  Day 11 - Non-Lesional | 53.37 [25.234 to 112.858] | 0.75 [0.257 to 2.208]
Statistical Analysis 1: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.488, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.395, 95% CI 2-sided [0.5429 to 3.5835] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.030, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.823, 95% CI 2-sided [1.1038 to 7.2210] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.127, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.077, 95% CI 2-sided [0.8122 to 5.3135] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.623, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.789, 95% CI 2-sided [0.3065 to 2.0331] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.328, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.627, 95% CI 2-sided [0.2450 to 1.6028] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.242, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.231, 95% CI 2-sided [0.5799 to 8.5866] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.321, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.977, 95% CI 2-sided [0.5137 to 7.6055] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.366, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.860, 95% CI 2-sided [0.4833 to 7.1564] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 9]; Test type: Superiority; p = 0.068, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.713, 95% CI 2-sided [0.9080 to 15.1856] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 10]; Test type: Superiority; p = 0.130, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.858, 95% CI 2-sided [0.7328 to 11.1434] — [estimate comment as in outcome 11, analysis 1]

14. Secondary Outcome: The Abundance of S. Aureus, as Measured by Culture, Between Treatment Groups on Lesional and Non-Lesional Skin Separately
Description: Amount of S. aureus present on lesional and non-lesional skin measured by Colony Forming Units per centimeter squared (CFU/cm^2)
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: CFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
CFU/cm^2
  Day 0 - Lesional | 3284.4 [1078.07 to 10006.32] | 1040.5 [221.94 to 4877.72]
  Day 0 - Non-lesional | 271.8 [91.38 to 808.34] | 112.4 [23.14 to 546.10]
  Day 4 - Lesional | 171.9 [56.44 to 523.85] | 2218.9 [473.30 to 10402.22]
  Day 4 - Non-lesional | 66.6 [22.39 to 198.07] | 644.1 [132.57 to 3128.93]
  Day 7 - Lesional | 301.7 [99.04 to 919.29] | 6716.4 [1432.67 to 31487.06]
  Day 7 - Non-lesional | 137.4 [46.21 to 408.78] | 1227.7 [252.71 to 5964.34]
  Day 8 - Lesional | 239.9 [77.90 to 738.56] | 2587.0 [518.99 to 12895.55]
  Day 8 - Non-lesional | 60.3 [20.06 to 181.16] | 649.8 [125.94 to 3352.62]
  Day 11 - Lesional | 81.8 [26.85 to 249.23] | 1856.5 [396.01 to 8703.40]
  Day 11 - Non-Lesional | 49.8 [16.75 to 148.19] | 135.1 [27.81 to 656.26]
Statistical Analysis 1: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Lesional Skin at Day 0 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.233, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.16, 95% CI 2-sided [0.476 to 20.952] — All reported statistics are back-transformed into the original units of measurement. Baseline is defined as the pre-dose value at treatment initiation/Day 0. TMT represents the numerator and Placebo the denominator
Statistical Analysis 2: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Lesional Skin at Day 4 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.008, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.08, 95% CI 2-sided [0.012 to 0.514] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Lesional Skin at Day 7 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.04, 95% CI 2-sided [0.007 to 0.298] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Lesional Skin at Day 8 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.017, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.09, 95% CI 2-sided [0.013 to 0.651] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Lesional Skin at Day 11 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.04, 95% CI 2-sided [0.007 to 0.292] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Non-lesional Skin at Day 0 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.358, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.42, 95% CI 2-sided [0.366 to 15.967] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Non-lesional Skin at Day 4 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.019, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.10, 95% CI 2-sided [0.016 to 0.683] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Non-lesional Skin at Day 7 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.023, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.11, 95% CI 2-sided [0.017 to 0.739] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Non-lesional Skin at Day 8 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.017, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.09, 95% CI 2-sided [0.013 to 0.647] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Non-lesional Skin at Day 11 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.299, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.37, 95% CI 2-sided [0.056 to 2.436] — [estimate comment as in outcome 14, analysis 1]

15. Secondary Outcome: The Abundance of S. Aureus, as Measured by qPCR (Quantitative Polymerase Chain Reaction), Between Treatment Groups on Lesional and Non-Lesional Skin Separately
Description: Amount of S. aureus present on lesional and non-lesional skin measured by relative Colony Forming Units per centimeter squared (rCFU/cm^2)
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: rCFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
rCFU/cm^2
  Day 0 - Lesional | 1177.8 [562.13 to 2467.96] | 788.3 [275.38 to 2256.52]
  Day 0 - Non-lesional | 319.8 [153.29 to 667.35] | 254.6 [88.61 to 731.38]
  Day 4 - Lesional | 839.3 [400.57 to 1758.66] | 950.3 [331.98 to 2720.26]
  Day 4 - Non-lesional | 347.3 [166.47 to 724.75] | 1091.1 [379.79 to 3134.70]
  Day 7 - Lesional | 1066.8 [509.11 to 2235.22] | 2696.7 [942.05 to 7719.32]
  Day 7 - Non-lesional | 604.5 [289.70 to 1261.22] | 745.5 [259.48 to 2141.71]
  Day 8 - Lesional | 915.3 [433.61 to 1931.94] | 2041.9 [661.92 to 6298.67]
  Day 8 - Non-lesional | 519.6 [247.14 to 1092.44] | 423.0 [140.27 to 1275.86]
  Day 11 - Lesional | 374.1 [178.56 to 783.96] | 791.0 [270.69 to 2311.43]
  Day 11 - Non-Lesional | 284.4 [136.31 to 593.45] | 361.4 [125.79 to 1038.27]
Statistical Analysis 1: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.538, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.49, 95% CI 2-sided [0.415 to 5.380]; All reported statistics are back-transformed into the original units of measurement. Baseline is defined as the pre-dose value at treatment initiation/Day 0. TMT represents the numerator and Placebo the denominator
Statistical Analysis 2: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p = 0.849, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.88, 95% CI 2-sided [0.245 to 3.180] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p = 0.155, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.40, 95% CI 2-sided [0.110 to 1.424] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p = 0.242, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.45, 95% CI 2-sided [0.117 to 1.722] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.258, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.47, 95% CI 2-sided [0.129 to 1.735] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 6]; Test type: Superiority; p = 0.726, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.26, 95% CI 2-sided [0.349 to 4.520] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 7]; Test type: Superiority; p = 0.080, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.32, 95% CI 2-sided [0.088 to 1.145] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 8]; Test type: Superiority; p = 0.748, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.81, 95% CI 2-sided [0.225 to 2.917] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 9]; Test type: Superiority; p = 0.760, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.23, 95% CI 2-sided [0.327 to 4.617] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 10]; Test type: Superiority; p = 0.713, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.79, 95% CI 2-sided [0.219 to 2.832] — [estimate comment as in outcome 14, analysis 1]

16. Secondary Outcome: The Abundance of S. Aureus, as Measured by Culture, Between Lesional and Non-Lesional Skin Within Each Treatment Group
Description: as for outcome 14
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: CFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
CFU/cm^2
  Day 0 - Lesional | 3284.4 [1078.07 to 10006.32] | 1040.5 [221.94 to 4877.72]
  Day 0 - Non-lesional | 271.8 [91.38 to 808.34] | 112.4 [23.14 to 546.10]
  Day 4 - Lesional | 171.9 [56.44 to 523.85] | 2218.9 [473.30 to 10402.22]
  Day 4 - Non-lesional | 66.6 [22.39 to 198.07] | 644.1 [132.57 to 3128.93]
  Day 7 - Lesional | 301.7 [99.04 to 919.29] | 6716.4 [1432.67 to 31487.06]
  Day 7 - Non-lesional | 137.4 [46.21 to 408.78] | 1227.7 [252.71 to 5964.34]
  Day 8 - Lesional | 239.9 [77.90 to 738.56] | 2587.0 [518.99 to 12895.55]
  Day 8 - Non-lesional | 60.3 [20.06 to 181.16] | 649.8 [125.94 to 3352.62]
  Day 11 - Lesional | 81.8 [26.85 to 249.23] | 1856.5 [396.01 to 8703.40]
  Day 11 - Non-Lesional | 49.8 [16.75 to 148.19] | 135.1 [27.81 to 656.26]
Statistical Analysis 1: Comparison: TMT Lotion; Lesional vs Non-Lesional within TMT at Day 0 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 12.08, 95% CI 2-sided [3.524 to 41.435] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: TMT Lotion; Lesional vs Non-Lesional within TMT at Day 4 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.131, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.58, 95% CI 2-sided [0.753 to 8.853] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion; Lesional vs Non-Lesional within TMT at Day 7 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.210, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.20, 95% CI 2-sided [0.640 to 7.527] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion; Lesional vs Non-Lesional within TMT at Day 8 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.031, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.98, 95% CI 2-sided [1.138 to 13.290] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion; Lesional vs Non-Lesional within TMT at Day 11 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.429, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.64, 95% CI 2-sided [0.479 to 5.630] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Placebo Lotion; Lesional vs Non-Lesional within Placebo at Day 0 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.010, Mixed Models Analysis; Geometric mean ratio (GMR) = 9.26, 95% CI 2-sided [1.712 to 50.043] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Placebo Lotion; Lesional vs Non-Lesional within Placebo at Day 4 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.150, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.45, 95% CI 2-sided [0.637 to 18.627] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Placebo Lotion; Lesional vs Non-Lesional within Placebo at Day 7 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.048, Mixed Models Analysis; Geometric mean ratio (GMR) = 5.47, 95% CI 2-sided [1.012 to 29.578] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Placebo Lotion; Lesional vs Non-Lesional within Placebo at Day 8 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.130, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.98, 95% CI 2-sided [0.665 to 23.821] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Placebo Lotion; Lesional vs Non-Lesional within Placebo at Day 11 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.002, Mixed Models Analysis; Geometric mean ratio (GMR) = 13.74, 95% CI 2-sided [2.542 to 74.304] — [estimate comment as in outcome 9, analysis 1]

17. Secondary Outcome: The Abundance of S. Aureus, as Measured by qPCR (Quantitative Polymerase Chain Reaction), Between Lesional and Non-Lesional Skin Within Each Treatment Group
Description: Amount of S.aureus present on lesional and non-lesional skin measured by relative Colony Forming Units per centimeter squared (rCFU/cm^2)
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: rCFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
rCFU/cm^2
  Day 0 - Lesional | 1177.8 [562.13 to 2467.96] | 788.3 [275.38 to 2256.52]
  Day 0 - Non-lesional | 319.8 [153.29 to 667.35] | 254.6 [88.61 to 731.38]
  Day 4 - Lesional | 839.3 [400.57 to 1758.66] | 950.3 [331.98 to 2720.26]
  Day 4 - Non-lesional | 347.3 [166.47 to 724.75] | 1091.1 [379.79 to 3134.70]
  Day 7 - Lesional | 1066.8 [509.11 to 2235.22] | 2696.7 [942.05 to 7719.32]
  Day 7 - Non-lesional | 604.5 [289.70 to 1261.22] | 745.5 [259.48 to 2141.71]
  Day 8 - Lesional | 915.3 [433.61 to 1931.94] | 2041.9 [661.92 to 6298.67]
  Day 8 - Non-lesional | 519.6 [247.14 to 1092.44] | 423.0 [140.27 to 1275.86]
  Day 11 - Lesional | 374.1 [178.56 to 783.96] | 791.0 [270.69 to 2311.43]
  Day 11 - Non-Lesional | 284.4 [136.31 to 593.45] | 361.4 [125.79 to 1038.27]
Statistical Analysis 1: Comparison: TMT Lotion; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.68, 95% CI 2-sided [1.689 to 8.028] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: TMT Lotion; [analysis description as in outcome 16, analysis 2]; Test type: Superiority; p = 0.027, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.42, 95% CI 2-sided [1.109 to 5.267] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion; [analysis description as in outcome 16, analysis 3]; Test type: Superiority; p = 0.153, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.76, 95% CI 2-sided [0.810 to 3.847] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion; [analysis description as in outcome 16, analysis 4]; Test type: Superiority; p = 0.160, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.76, 95% CI 2-sided [0.799 to 3.884] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion; [analysis description as in outcome 16, analysis 5]; Test type: Superiority; p = 0.489, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.32, 95% CI 2-sided [0.603 to 2.868] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Placebo Lotion; [analysis description as in outcome 16, analysis 6]; Test type: Superiority; p = 0.044, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.10, 95% CI 2-sided [1.032 to 9.295] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Placebo Lotion; [analysis description as in outcome 16, analysis 7]; Test type: Superiority; p = 0.805, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.87, 95% CI 2-sided [0.290 to 2.614] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Placebo Lotion; [analysis description as in outcome 16, analysis 8]; Test type: Superiority; p = 0.022, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.62, 95% CI 2-sided [1.205 to 10.859] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Placebo Lotion; [analysis description as in outcome 16, analysis 9]; Test type: Superiority; p = 0.010, Mixed Models Analysis; Geometric mean ratio (GMR) = 4.83, 95% CI 2-sided [1.458 to 15.978] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Placebo Lotion; [analysis description as in outcome 16, analysis 10]; Test type: Superiority; p = 0.169, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.19, 95% CI 2-sided [0.716 to 6.692] — [estimate comment as in outcome 9, analysis 1]

18. Secondary Outcome: The Change From Baseline Levels of S. Aureus Abundance, as Measured by Culture, Between Lesional and Non-Lesional Skin Within Each Treatment Group
Description: as for outcome 14
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: CFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
CFU/cm^2
  Day 0 - Lesional | 0.12 [0.039 to 0.380] | 0.44 [0.085 to 2.248]
  Day 0 - Non-lesional | 0.69 [0.221 to 2.161] | 1.45 [0.282 to 7.442]
  Day 4 - Lesional | 0.05 [0.017 to 0.164] | 2.13 [0.415 to 10.964]
  Day 4 - Non-lesional | 0.25 [0.078 to 0.767] | 5.73 [1.114 to 29.455]
  Day 7 - Lesional | 0.09 [0.029 to 0.288] | 6.46 [1.256 to 33.186]
  Day 7 - Non-lesional | 0.51 [0.162 to 1.583] | 10.92 [2.124 to 56.147]
  Day 8 - Lesional | 0.07 [0.023 to 0.231] | 2.49 [0.456 to 13.546]
  Day 8 - Non-lesional | 0.22 [0.070 to 0.700] | 5.78 [1.061 to 31.493]
  Day 11 - Lesional | 0.02 [0.008 to 0.078] | 1.78 [0.347 to 9.173]
  Day 11 - Non-Lesional | 0.18 [0.059 to 0.574] | 1.20 [0.234 to 6.178]
Statistical Analysis 1: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.035, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.176, 95% CI 2-sided [0.0351 to 0.8807] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.060, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.214, 95% CI 2-sided [0.0427 to 1.0702] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.038, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.182, 95% CI 2-sided [0.0363 to 0.9100] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.179, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.329, 95% CI 2-sided [0.0650 to 1.6691] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.015, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.136, 95% CI 2-sided [0.0271 to 0.6805] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.309, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.302, 95% CI 2-sided [0.0299 to 3.0493] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.401, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.372, 95% CI 2-sided [0.0369 to 3.7569] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.655, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.591, 95% CI 2-sided [0.0586 to 5.9658] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 9]; Test type: Superiority; p = 0.488, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.430, 95% CI 2-sided [0.0395 to 4.6836] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 10]; Test type: Superiority; p = 0.737, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.485, 95% CI 2-sided [0.1471 to 14.9869] — [estimate comment as in outcome 11, analysis 1]

19. Secondary Outcome: The Change From Baseline Levels of S. Aureus Abundance, as Measured by qPCR (Quantitative Polymerase Chain Reaction), Between Lesional and Non-Lesional Skin Within Each Treatment Group
Description: as for outcome 15
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: rCFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
rCFU/cm^2
  Day 0 - Lesional | 0.72 [0.314 to 1.637] | 0.55 [0.170 to 1.814]
  Day 0 - Non-lesional | 2.89 [1.258 to 6.646] | 1.11 [0.341 to 3.645]
  Day 4 - Lesional | 0.71 [0.312 to 1.628] | 1.21 [0.369 to 3.943]
  Day 4 - Non-lesional | 1.09 [0.475 to 2.480] | 4.29 [1.310 to 14.020]
  Day 7 - Lesional | 0.91 [0.397 to 2.069] | 3.42 [1.046 to 11.190]
  Day 7 - Non-lesional | 1.89 [0.827 to 4.317] | 2.93 [0.895 to 9.579]
  Day 8 - Lesional | 0.78 [0.338 to 1.787] | 2.59 [0.741 to 9.051]
  Day 8 - Non-lesional | 1.62 [0.707 to 3.735] | 1.66 [0.487 to 5.671]
  Day 11 - Lesional | 0.32 [0.139 to 0.726] | 1.00 [0.301 to 3.346]
  Day 11 - Non-Lesional | 0.89 [0.389 to 2.031] | 1.42 [0.434 to 4.644]
Statistical Analysis 1: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.011, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.248, 95% CI 2-sided [0.0844 to 0.7281] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.440, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.656, 95% CI 2-sided [0.2245 to 1.9178] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.178, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.479, 95% CI 2-sided [0.1640 to 1.4007] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.180, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.478, 95% CI 2-sided [0.1624 to 1.4091] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.060, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.357, 95% CI 2-sided [0.1222 to 1.0441] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.373, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.498, 95% CI 2-sided [0.1068 to 2.3188] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.106, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.281, 95% CI 2-sided [0.0604 to 1.3106] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.843, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.168, 95% CI 2-sided [0.2507 to 5.4434] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 9]; Test type: Superiority; p = 0.587, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.559, 95% CI 2-sided [0.3122 to 7.7818] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Placebo Lotion; [analysis description as in outcome 9, analysis 10]; Test type: Superiority; p = 0.661, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.707, 95% CI 2-sided [0.1495 to 3.3426] — [estimate comment as in outcome 11, analysis 1]

20. Secondary Outcome: The Abundance of Bacterial Deoxyribonucleic Acid (DNA) of Combined S. Hominis, as Measured by Quantitative Polymerase Chain Reaction (qPCR), Between Treatment Groups on Lesional and Non-Lesional Skin Separately
Description: Amount of combined S. hominis present on lesional and non-lesional skin measured by relative Colony Forming Units per centimeter squared (rCFU/cm^2)
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: rCFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
rCFU/cm^2
  Day 0 (post-treatment) - Lesional | 103291.5 [64503.91 to 165387.54] | 86.3 [43.92 to 169.52]
  Day 0 (post-treatment) - Non-lesional | 82176.8 [50998.80 to 132415.39] | 108.5 [55.21 to 213.23]
  Day 4 - Lesional | 97810.2 [61086.59 to 156610.99] | 125.5 [63.89 to 246.61]
  Day 4 - Non-lesional | 40682.3 [25406.91 to 65141.85] | 203.7 [103.65 to 400.33]
  Day 7 - Lesional | 98401.7 [61456.00 to 157558.06] | 146.1 [74.36 to 287.03]
  Day 7 - Non-lesional | 46775.4 [29212.14 to 74898.23] | 92.0 [46.81 to 180.79]
  Day 8 - Lesional | 6068.6 [3765.70 to 97793.98] | 100.9 [48.16 to 211.61]
  Day 8 - Non-lesional | 9675.2 [6003.60 to 15592.22] | 89.7 [43.79 to 183.75]
  Day 11 - Lesional | 743.8 [464.54 to 1190.97] | 196.4 [98.05 to 393.42]
  Day 11 - Non-Lesional | 1081.7 [675.56 to 1732.08] | 67.2 [34.22 to 132.16]
Statistical Analysis 1: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Lesional Skin at Day 0 (post-treatment) A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 1197.16, 95% CI 2-sided [525.563 to 2726.953] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 779.24, 95% CI 2-sided [342.093 to 1774.996] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 673.56, 95% CI 2-sided [295.697 to 1534.265] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 60.12, 95% CI 2-sided [24.920 to 145.027]; [other analysis details as in outcome 15, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.002, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.79, 95% CI 2-sided [1.636 to 8.767] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Non-lesional Skin at Day 0 (post-treatment) A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and lesional swab status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 757.38, 95% CI 2-sided [331.143 to 1732.242] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 7]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 199.71, 95% CI 2-sided [87.636 to 455.127] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 8]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 508.45, 95% CI 2-sided [223.113 to 1158.715]; [other analysis details as in outcome 15, analysis 1]
Statistical Analysis 9: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 9]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 107.86, 95% CI 2-sided [45.568 to 255.313] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 10]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 16.09, 95% CI 2-sided [7.058 to 36.657] — [estimate comment as in outcome 14, analysis 1]

21. Secondary Outcome: The Abundance of Bacterial Deoxyribonucleic Acid (DNA) of Combined Staphylococci, as Measured by qPCR (Quantitative Polymerase Chain Reaction), Between Treatment Groups on Lesional and Non-Lesional Skin Separately
Description: Amount of combined Staphylococci present on lesional and non-lesional skin measured by relative Colony Forming Units per centimeter squared (rCFU/cm^2)
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: rCFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
rCFU/cm^2
  Day 0 (post-treatment) - Lesional | 169474.3 [101234.39 to 283713.19] | 1186.0 [569.89 to 2468.35]
  Day 0 (post-treatment) - Non-lesional | 201324.3 [119927.33 to 337966.84] | 754.4 [361.30 to 1575.17]
  Day 4 - Lesional | 144236.8 [86158.92 to 241463.63] | 4099.1 [1969.61 to 8530.96]
  Day 4 - Non-lesional | 111784.4 [67001.83 to 186498.58] | 2188.7 [1048.21 to 4569.94]
  Day 7 - Lesional | 171843.8 [102649.79 to 287679.90] | 4126.8 [1982.93 to 8588.65]
  Day 7 - Non-lesional | 101610.2 [60903.58 to 169524.19] | 1355.5 [649.17 to 2830.24]
  Day 8 - Lesional | 15115.6 [8972.04 to 25466.03] | 4190.4 [1885.57 to 9312.50]
  Day 8 - Non-lesional | 23330.8 [13891.98 to 39182.93] | 895.4 [410.93 to 1950.87]
  Day 11 - Lesional | 2874.3 [1716.97 to 4811.87] | 2063.5 [973.77 to 4372.86]
  Day 11 - Non-Lesional | 3135.3 [1879.25 to 5230.87] | 918.6 [439.96 to 1918.12]
Statistical Analysis 1: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 142.89, 95% CI 2-sided [58.484 to 349.119] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 35.19, 95% CI 2-sided [14.402 to 85.972] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 41.64, 95% CI 2-sided [17.043 to 101.739] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p = 0.008, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.61, 95% CI 2-sided [1.395 to 9.330] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.474, Mixed Models Analysis; Geometric mean ratio (GMR) = 1.39, 95% CI 2-sided [0.561 to 3.458] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 20, analysis 6]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 266.87, 95% CI 2-sided [108.860 to 654.231] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 7]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 51.07, 95% CI 2-sided [20.907 to 124.768] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Non-lesional Skin at Day 7 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 74.96, 95% CI 2-sided [30.686 to 183.125] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: TMT Lotion; TMT vs Placebo on Non-lesional Skin at Day 8 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 26.06, 95% CI 2-sided [10.262 to 66.169] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: TMT Lotion vs Placebo Lotion; TMT vs Placebo on Non-lesional Skin at Day 11 A random effects linear model with the log10 transformed numeric response variable was used, adjusting for treatment group, baseline value, site, lesional swab status, and study day, in addition to all pairwise interactions between day, group and status and a 3-way interaction. Random effects of subject and time point nested within subject were also included in the model; Test type: Superiority; p = 0.007, Mixed Models Analysis; Geometric mean ratio (GMR) = 3.41, 95% CI 2-sided [1.397 to 8.338] — [estimate comment as in outcome 14, analysis 1]

22. Secondary Outcome: The Abundance of Combined Bacterial Deoxyribonucleic Acid (DNA), as Measured by qPCR (Quantitative Polymerase Chain Reaction), Between Treatment Groups on Lesional and Non-Lesional Skin Separately
Description: Amount of combined bacteria present on lesional and non-lesional skin measured by relative Colony Forming Units per centimeter squared (rCFU/cm^2)
Time Frame: Days 0 (1 hour post treatment), 4, 7, 8 and 11
Population: as for outcome 5
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: rCFU/cm^2
Arm/Group | TMT Lotion | Placebo Lotion
Number analyzed (Participants) | 35 | 17
rCFU/cm^2
  Day 0 (post-treatment) - Lesional | 42609.4 [26067.18 to 69649.16] | 833.8 [412.72 to 1684.66]
  Day 0 (post-treatment) - Non-lesional | 45142.5 [27483.01 to 74149.34] | 812.9 [401.98 to 1643.95]
  Day 4 - Lesional | 37621.5 [23015.76 to 61496.03] | 2923.3 [1446.93 to 5906.17]
  Day 4 - Non-lesional | 19461.7 [11918.85 to 31777.91] | 1652.0 [816.90 to 3340.83]
  Day 7 - Lesional | 37338.7 [22842.73 to 61033.73] | 3259.5 [1613.31 to 6585.30]
  Day 7 - Non-lesional | 25114.3 [15380.71 to 41007.86] | 1084.1 [536.08 to 2192.36]
  Day 8 - Lesional | 5072.8 [3083.69 to 8345.12] | 2097.8 [974.26 to 4517.19]
  Day 8 - Non-lesional | 6323.9 [3848.09 to 10392.63] | 572.1 [271.26 to 1206.67]
  Day 11 - Lesional | 1204.9 [737.15 to 1969.6] | 1596.9 [776.65 to 3283.46]
  Day 11 - Non-Lesional | 1666.8 [1020.81 to 2721.67] | 686.1 [339.26 to 1387.44]
Statistical Analysis 1: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 51.10, 95% CI 2-sided [21.692 to 120.379] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 12.87, 95% CI 2-sided [5.463 to 30.317] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 11.46, 95% CI 2-sided [4.863 to 26.986] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p = 0.058, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.42, 95% CI 2-sided [0.971 to 6.024] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.526, Mixed Models Analysis; Geometric mean ratio (GMR) = 0.75, 95% CI 2-sided [0.315 to 1.805] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 20, analysis 6]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 55.53, 95% CI 2-sided [23.490 to 131.279] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 7]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 11.78, 95% CI 2-sided [5.000 to 27.755] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 8]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 23.17, 95% CI 2-sided [9.833 to 54.579] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 9]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric mean ratio (GMR) = 11.05, 95% CI 2-sided [4.516 to 27.052] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: TMT Lotion vs Placebo Lotion; [analysis description as in outcome 14, analysis 10]; Test type: Superiority; p = 0.042, Mixed Models Analysis; Geometric mean ratio (GMR) = 2.43, 95% CI 2-sided [1.031 to 5.724] — [estimate comment as in outcome 14, analysis 1]

ADVERSE EVENTS:
Time Frame: 8 days
Description: Adverse Events (AEs) grade 1 or higher.
  Graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Arm/Group | Targeted Microbiome Transplant (TMT) | Placebo Lotion
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/18
Other Adverse Events (participants affected / at risk) | 21/36 | 16/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted Microbiome Transplant (TMT) (N=36) | Placebo Lotion (N=18)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 8 (14) | 4 (11)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (21) | 7 (18)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 15 (28) | 11 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03151148/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03151148/SAP_001.pdf